CLINICAL TRIAL: NCT03999151
Title: A Randomized Controlled Trial of Diet & Exercise Interventions Among Men With Prostate Cancer - II (Prostate 8-II)
Brief Title: Diet and Exercise Interventions Among Men With Prostate Cancer (Prostate 8-II)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 175513-HDFCCC; NCI-2018-02347 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 5R01CA207749-05 (NIH)
Record Dates: First submitted 2019-06-21; First posted 2019-06-26 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Exercise; Diet; Lifestyle; Digital; Text messaging; Coach
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A: Reference Group (Active Comparator): Arm A will receive print educational materials about the benefits of exercise and diet for men with prostate cancer, with recommendations geared at men living with prostate cancer, mailed around the date of surgery. They also receive a 10-week text messaging program focused on recovery after radical prostatectomy surgery.
  Interventions: Behavioral: Exercise and Diet
- Arm B (Arm A + Exercise) (Experimental): Arm B receives the following: Arm A material plus access to an online portal with additional educational materials to help improve exercise habits and various tools, such as the ability to track exercise; additional educational print materials on exercise; additional text messages over 2 years that supports healthy exercise habits; and a 1-hour phone session at the start of the study followed by eight 30-minute quarterly phone sessions with an exercise coach over 2 years.
  Interventions: Behavioral: Exercise and Diet
- Arm C (Arm A + Diet) (Experimental): Arm C receives the following: Arm A material plus access to an online portal with additional educational materials to help improve diet habits and various tools, such as the ability to track diet; additional educational print materials on diet; additional text messages over 2 years that supports healthy diet habits; and a 1-hour phone session at the start of the study followed by eight 30-minute quarterly phone sessions with a diet coach over 2 years.
  Interventions: Behavioral: Exercise and Diet
- Arm D (Arm A + Exercise + Diet) (Experimental): Arm D receives the following: Arm A material plus access to an online portal with additional educational materials to help improve exercise and diet habits and various tools, such as the ability to track exercise and diet; additional educational print materials on exercise and diet; additional text messages over 2 years that supports healthy exercise and diet habits; a 1-hour phone session at the start of the study followed by eight 30-minute quarterly phone sessions with an exercise coach over 2 years; and a 1-hour phone session at the start of the study followed by eight 30-minute quarterly phone sessions with a diet coach over 2 years.
  Interventions: Behavioral: Exercise and Diet

INTERVENTIONS:
Behavioral: Exercise and Diet — Behavioral program provides access to educational materials + clinical texting program (Arm A) + participant portal, text messaging, and coaching (Arms B-D)

SUMMARY:
The Prostate 8-II study is a randomized controlled trial of testing different combinations of educational and supportive tools related to diet and exercise to evaluate biological, clinical, and quality of life outcomes in men choosing radical prostatectomy as treatment for prostate cancer.

DETAILED DESCRIPTION:
This is a PI initiated, randomized controlled trial of four exercise and diet interventions among men opting for radical prostatectomy for prostate cancer.

The Prostate 8-II study enrolls men up to 8 weeks prior to surgery and participants remain on study for 24 cycles after surgery (1 cycle=28 days). After obtaining written informed consent, enrolled subjects will be scheduled for the baseline assessments. All participants will receive Group A educational materials and tools, but these will be distributed at different times based on group assignment. The other 3 groups will receive different combinations of exercise (Group B), diet (Group C) and exercise and diet (Group D) tools. Men in all arms will be asked to complete questionnaires at baseline, pre-surgery, and at cycles 6,12, & 24 post-surgery, and complete blood and urine collection, diet recall, and accelerometer measurement at select time points. Specimens from biopsy and radical prostatectomy will be reviewed by the investigators' collaborator, GenomeDx, for RNA characterization and assessment of the genomic risk scores. Participants will be followed for 30 days after completion of the 2-year 24-cycle intervention period or removal from the study, or until death, whichever occurs first for any treatment-related adverse events. Following the completion of the intervention, participant's treatment and disease status will be collected on a yearly basis, for 3 more years.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years
2. Diagnosed with non-metastatic prostate cancer and choose radical prostatectomy (RP) as primary treatment.
3. Able to speak and read English
4. Regular access to the Internet (via a computer, tablet, or phone) and text messaging capabilities on the phone
5. Ability to understand a written informed consent document, and the willingness to sign it

Exclusion Criteria:

1. Cannot have neoadjuvant radiation or hormone therapy planned at time of enrollment (if enrolling >4 weeks prior to RP).
2. Men who have contraindications to exercise based the American College of Sports Medicine 2016 Exercise pre-participation screening criteria (https://www.ncbi.nlm.nih.gov/pubmed/26473759), and who do not receive a physician clearance to participate in the moderate to vigorous intensity physical activity with one or more of the following self-reported conditions:

   1. Heart attack
   2. Heart surgery, cardiac catheterization, or coronary angioplasty
   3. Pacemaker/implantable cardiac defibrillator/rhythm disturbance
   4. Heart valve disease
   5. Heart failure
   6. Heart transplantation
   7. Congenital heart disease
   8. Diabetes
   9. Kidney (renal) disease
   10. Chest discomfort with exertion
   11. Unreasonable breathlessness
   12. Dizziness, fainting, or blackouts
   13. Ankle swelling
   14. Unpleasant awareness of forceful, rapid or irregular heart rate
   15. Burning or cramping sensations in your lower legs when walking short distance
3. Men already meeting aerobic AND resistance exercise recommendations. To be eligible, must not meet at least one of the following: (1) 150 minutes per week of planned moderate aerobic exercise or 75 minutes per week of planned vigorous aerobic exercise or combination;(2) Two or more days per week of resistance exercise; (3) Eight or more resistance exercises per session
4. Men who are already meeting all of the 7 prostate-specific dietary recommendations

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with detectable levels of Prostate-specific antigen (PSA) | 6 months and 24 months post-surgery
  Detectable PSA will be defined based on current practice at the time of analysis. Point estimate and 95% confidence interval of the proportion of detectable PSA at 6 months and 2 years post-surgery for each group will be reported. In addition, Pearson's Chi-square test will be used to test if there are differences in the proportion of detectable PSA at least 6 weeks post-surgery among the groups. If there is a significant difference observed, a 2-sample proportion test to compare Groups B, C, and D, separately, with Group A and one another for each post-intervention time point will be performed. Point estimates and 95% confidence intervals of the recurrence proportion will be obtained for each group
Annual PSA recurrence rate | Up to 5 years
  Risk of cancer recurrence (based on current practice) measured using standard criteria using a log- rank test to evaluate the time to recurrence among groups, and multivariate Cox proportional hazards regression to obtain a hazard ratio for the time to recurrence

SECONDARY OUTCOMES:
Changes in Messenger Ribonucleic Acid (mRNA) expression patterns (focusing on change between biopsy and RP) | From baseline to up to 8 weeks
  Effect of intervention on changes in mRNA expression patterns using the 1.4 million marker Affymetrix 1.0 Human Exon Array, in formalin-fixed paraffin-embedded (FFPE) prostate biopsy and prostatectomy tissue to determine which genes are differentially expressed from biopsy to RP within each group. If the expression is significantly different in at least one of the groups, the change of RNA expression level will be compared among all groups by ANOVA. If there is a significant difference observed, we will perform pairwise comparisons among the groups. Multiple testing adjustment will be done by controlling false discovery rate
Decipher score (focusing on change between biopsy and RP) | From baseline to up to 8 weeks
  Assessment of genomic classifiers, using the 1.4 million marker Affymetrix 1.0 Human Exon Array, in FFPE (formalin-fixed paraffin embedded) prostate biopsy and radical prostatectomy tissue. Each score ranges from 0 to 100 and can be interpreted as a probability of progression. The 2-sample proportion test will be used to compare the proportion of reduction in the genomic score between Groups B, C, and D, separately with Group A first. Significant mean changes in the Decipher score will be tested using Analysis of Variance (ANOVA). If there is a significant difference observed, pairwise comparisons among the groups will be performed. A regression model will be built using an indicator for group and stratification factors such as age at diagnosis and surgical parameters (e.g., CAPRA-S) which have been determined to be potential covariates.
Change in sexual function as measured by the Expanded Prostate Cancer Index Composite Short Form (EPIC-26) | Baseline, and 6 months, 12 months, and 24 months post-surgery
  The EPIC-26 will be used to determine the impact of quality of life issues on the sexual function domain. Response options for each EPIC item form a Likert scale, and the raw score of each item is then transformed linearly to a 0-100 scale. Multiple items are combined and then averaged to form the domain scores and total score at each time point also ranging from 0-100, with higher scores representing better health related quality of life (HRQOL).
Change in urinary function as measured by the EPIC-26 | Baseline, and 6 months, 12 months, and 24 months post-surgery
  The EPIC-26 will be used to determine the impact of quality of life issues on the urinary function domain. Response options for each EPIC item form a Likert scale, and the raw score of each item is then transformed linearly to a 0-100 scale. Multiple items are combined and then averaged to form the domain scores and total score at each time point also ranging from 0-100, with higher scores representing better health related quality of life (HRQOL).
Change in scores on the general anxiety scale of the Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline, and 6 months, 12 months, and 24 months post-surgery
  General anxiety items usually has five response options ranging in value from one to five with a higher value indicating a greater degree of anxiety. The total raw score is the sum the values of the response to each question, and then converted to a scaled T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10.
Change in scores on the Memorial Anxiety Scale for Prostate Cancer (MAX-PC) | Baseline, and 6 months, 12 months, and 24 months post-surgery
  Memorial Anxiety Scale for Prostate Cancer (MAX-PC) - 18 items assessing prostate cancer anxiety, PSA anxiety, and fear of recurrence; range 0-54; smaller number is better.
Change in scores on the general depression scale of the Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline, and 6 months, 12 months, and 24 months post-surgery
  General depression items usually has five response options ranging in value from one to five with a higher value indicating a greater degree of depression. The total raw score is the sum the values of the response to each question, and then converted to a scaled T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10.
Change in scores on the SF-12 | Baseline, and 6 months, 12 months, and 24 months post-surgery
  The SF-12 is a 12-item questionnaire used to assess generic health outcomes from the patient's perspective. The SF-12 consists of a subset of 12 items from the SF-36® Health Survey (SF-36) and measures two composite outcomes assessing mental health composite score (MCS) and physical health composite scores (PCS). The PCS & MCS are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. The absolute change in item score by group from baseline up to 12 months was used to assess the quality of life/psychosocial impact on the patients with a larger scores indicating a greater degree of change on physical and mental health.
Change in physical activity over time | Baseline, and 6 months, 12 months, and 24 months post-surgery
  Patients will wear an Actigraph GT3X+ accelerometer on their wrist for 7 consecutive days to measure physical activity
Change in scores on the Godin-Shephard Leisure-Time Physical Activity Questionnaire | Baseline, and 6 months, 12 months, and 24 months post-surgery
  The Godin-Shephard Leisure-Time Physical Activity Questionnaire measures the frequency and duration of various types of physical activity (strenuous, moderate, light) and each is weighted by multiplying the frequency by a corresponding multiplier (x9, x5, x3 respectively) during a typical 7-Day period. The weekly leisure activity score = (9 × Strenuous) + (5 × Moderate) + (3 × Light). A score of 24 units or more indicates a status of "Active", 14 - 23 units "Moderately Active" and < 14 units "Insufficiently Active/Sedentary".
Change in Harvard Food Frequency Questionnaire (FFQ) over time | Baseline, and 6 months, 12 months, and 24 months post-surgery
  The FFQ is a self-administered questionnaire to assess intake of various nutrients. Nutrient intakes are computed by assigning a daily frequency weight
Diet recall | Baseline, and 6 months, 12 months, and 24 months post-surgery
  Two online 24-hour diet recalls as recommended by the National Cancer Institute's Diet Assessment Primer
Intervention feasibility and acceptability (intervention arms) | Baseline, and 6 months, 12 months, and 24 months post-surgery
  Various metrics for study feasibility (e.g., text message, portal, and coaching use) will be measured over time. Study acceptability will be evaluated by survey and in a subset, by phone interview. Descriptive data of these metrics across arms will be reported
Self/efficacy confidence in adopting healthy behaviors over time | Baseline, and 6 months, 12 months, and 24 months post-surgery
  Confidence scores in adopting dietary and physical activity behaviors at for each group using descriptive statistics, such as means, medians, and interquartile range will be reported using descriptive statistics.
Changes in scores on the Pittsburgh Sleep Quality Index (PSQI) | Baseline, and 6 months, 12 months, and 24 months post-surgery
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality
Changes in perceived social support | Baseline, and 6 months, 12 months, and 24 months post-surgery
  Social support will be measured using published measures from University of California, San Diego (http://sallis.ucsd.edu/measure_socialsupport.html

CONTACTS AND LOCATIONS:
Overall Officials: Stacey A Kenfield, DSc, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco (UCSF), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT03999151/ICF_000.pdf